CLINICAL TRIAL: NCT02207868
Title: 3D Echo Evaluation of the Ventricles in Sclero Associated Severe PAH (EVA 3D Pilot Study)
Brief Title: 3D Echo Evaluation of the Ventricles in Sclero Associated Severe PAH
Acronym: EVA3D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Steringer-Mascherbauer (Other)
Responsible Party: Sponsor-Investigator, Regina Steringer-Mascherbauer, OA Dr., Elisabethinen Hospital
Organization: Elisabethinen Hospital (Other)
Other Study IDs: EVA 3D
Record Dates: First submitted 2014-07-21; First posted 2014-08-04 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment

SUMMARY:
The aim of the study is to document the left and right ventricular function in patients with sclerodermia associated pulmonal arterial hypertension via 3D echocardiography. The results of this study should help to generate hypothesis for further future studies.

The primary hypothesis is that the increased use of modern image guided methods could provide essential aspects for the follow up.

DETAILED DESCRIPTION:
The 3D echocardiography could provide early and detailed information about the changes in the left and right ventricle.

The prediction of sclerodermia associated pulmonary arterial hypertension (PAH) is rather adverse, so it makes sense to evaluate relevant changes of the left-ventricular longitudinal strain soon to adapt the PAH specific therapy accordingly.

ELIGIBILITY:
Inclusion Criteria:

* age >17
* pulmonary arterial hypertension (PAH) associated with WHO group 1 who start a parenteral prostanoid-therapy
* written informed consent
* prostanoid naive
* no change of the PAH specific therapy within 3 weeks of the recruitment to the study

Exclusion Criteria:

* pregnancy and lactation period
* Women of child bearing potential who do not use an effective and secure method for birth control
* severe chronic kidney insufficiency (glomerular filtration rate <30), which will remain for more than 3 months
* liver-insufficiency Child C
* life expectancy shorter than the course of the study (for example because of malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pulmonary arterial hypertension associated with WHO group 1 who start with a parenteral prostanoidtherapy.
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change of the left ventricular longitudinal strain | day 90 (+/- 7 days)
  echocardiography

SECONDARY OUTCOMES:
wall thickness | 90 days (+/- 7 days)
  echocardiography
left ventricular ejection fracture | 90 days (+/- 7 Days)
  echocardiography
left ventricular stroke volume | 90 days (+/- 7 days)
  echocardiography
Tricuspid Annular Plane Systolic Excursion (TAPSE) | 90 days (+/- 7 days)
  echocardiography
right ventricular fractional area change | 90 (+/- 7 days)
  echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Regina Steringer-Mascherbauer, MD, Principal Investigator — Krankenhaus der Elisabethinen Linz GmbH
Locations (1):
- Krankenhaus der Elisabethinen Linz GmbH, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided